CLINICAL TRIAL: NCT01107834
Title: Left Ventricular Function in HIV-Negative Children Exposed to HIV and HAART In Utero
Brief Title: Heart Function in HIV-Negative Children Exposed to HIV and HAART
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, W. Todd Cade, Assistant Professor of Physical Therapy and Medicine, Washington University School of Medicine
Other Study IDs: 10-0121
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Results first posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-06

CONDITIONS: HIV Infections
Keywords: HIV; heart function; HAART; in utero; children
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Control: HIV-negative children born to healthy, HIV-negative women
- Exposed to HIV/HAART: HIV-negative children exposed to HIV and HAART in utero

SUMMARY:
HIV-uninfected children born to HIV+ women have low level heart problems at birth which may predispose them to heart failure, arrythmias and heart attack later in life. The impact of these heart problems on future heart health is unclear as it is unknown if heart problems in these children persist, worsen or resolve in pre-pubescence. The objective of this study is to characterize heart function in HIV-negative pre-pubertal children born to HIV+ women and exposed to HIV and HAART in utero and compare them to age and gender matched healthy children born to HIV-negative women. Through this objective we will determine if heart problems in HIV-negative children born to HIV+ women and exposed to HAART in utero persists, worsens, or resolves during pre-pubescence.

DETAILED DESCRIPTION:
Significance:

Approximately 700,000 children annually are born to HIV-infected mothers throughout the world, but with the advent of perinatal highly active antiretroviral therapy (HAART), the majority of children are born uninfected in Westernized nations and those uninfected are increasing in developing nations. Uninfected children exposed to HIV and HAART in utero, have subclinical left ventricular dysfunction (LVD) at birth which may predispose them to heart failure, conduction abnormalities and myocardial infarction later in life. The impact of this LVD on future cardiac risk is unclear as it is unknown if LVD in these children persist, worsen or resolve in pre-pubescence.

Study objectives:

The objective of this study is to characterize left ventricular function in HIV-negative pre-pubertal children born to HIV+ women and exposed to HIV and HAART in utero and compare them to age and gender matched healthy children born to HIV-negative women. Through this objective we will determine if LVD in HIV-negative children born to HIV+ women and exposed to HAART in utero persists, worsens, or resolves during pre-pubescence. If LVD persists or worsens in pre-pubescence, these data will lead to future studies examining mechanisms of and treatments for LVD in these children and will significantly impact the clinical monitoring and care of these children. If LVD resolves during pre-pubescence, then these data will provide important information that clinical cardiac monitoring may not be critical in this population.

Methods:

We plan to examine left ventricular function in 30 HIV-negative children born to HIV+ women and exposed to HAART in utero and compare them to 30 healthy age and gender matched children born to HIV-negative women. Left ventricular function will be examined by 2-D, Doppler and Tissue Doppler imaging echocardiography using a General Electric Vivid 7® ultrasound machine. Left ventricular measures will include left ventricular structure and dimensions, systolic and diastolic flow rates, wall velocities during systole and diastole and systolic and diastolic strain and strain rates (sensitive measures of myocardial contractility). Echocardiographic measures will take place in the Cardiovascular Imaging Laboratory (CVIL) at Washington University School of Medicine by a certified cardiac ultrasonographer and data will be processed, analyzed and interpreted by the ultrasonographer, a consulting cardiologist and the principal investigator.

Outcomes:

Primary outcomes will include measures of left ventricular function: left ventricular mass, left ventricular end diastolic dimension, fractional shortening, systolic and diastolic wall velocities (tissue Doppler imaging) and systolic and diastolic strain and strain rates (2-D speckle tracking methodology).

ELIGIBILITY:
Inclusion Criteria:

1. Age 5-12 years
2. Tanner stage I-III
3. Born to HIV+ mother
4. No HIV infection
5. Had taken standard of care prophylactic HAART at birth-1 month of age
6. Child currently not taking medications or have medical diagnosis that would affect left ventricular function
7. Mother was taking HAART during pregnancy (standard of care)
8. Mother was not using illegal drugs during pregnancy
9. No intrauterine growth restriction diagnosis during pregnancy
10. During pregnancy, mother will not have a diagnosis of type 2 diabetes or gestational diabetes.

Exclusion Criteria:

1. Age 5-12 years
2. Tanner stage I-III
3. Born to HIV-negative mother
4. Mother was not a frequent exerciser during pregnancy (>2x/week)
5. Mother will not have gestational diabetes or a diagnosis of type 2 diabetes during pregnancy of the child being studied
6. Child currently not taking medications or have medical diagnosis that would affect left ventricular function

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: HIV-negative children will be recruited through their HIV+ mothers who are seen at the AIDS Clinical Trials Unit at Washington University and surrounding St. Louis community clinics. HIV-negative children will be recruit through Washington University and surrounding St. Louis pediatric clinics, and through Washington University Volunteers for Health service.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T Cade, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Cade WT, Waggoner AD, Hubert S, Krauss MJ, Singh GK, Overton ET. Reduced diastolic function and left ventricular mass in HIV-negative preadolescent children exposed to antiretroviral therapy in utero. AIDS. 2012 Oct 23;26(16):2053-8. doi: 10.1097/QAD.0b013e328358d4d7. PMID 22874520

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Control | Exposed to HIV/HAART
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Exposed to HIV/HAART | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 8 (2) | 8 (3) | 8 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 19 | 19 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 23 | 45
  White | 6 | 6 | 12
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Mass Index
Description: left ventricular mass index measured by 2D echocardiography
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: g/m2
Arm/Group | Healthy Control | Exposed to HIV/HAART
Number analyzed (Participants) | 30 | 30
g/m2 | 67 (12) | 60 (9)
Statistical Analysis 1: Comparison: Healthy Control vs Exposed to HIV/HAART; T-test to detect differences between groups; Test type: Superiority or Other; p = 0.27, t-test, 2 sided

2. Primary Outcome: Fractional Shortening
Description: Fractional shortening measured by M-mode cardiography
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of full contraction
Arm/Group | Healthy Control | Exposed to HIV/HAART
Number analyzed (Participants) | 30 | 30
percentage of full contraction | 36 (5) | 37 (7)
Statistical Analysis 1: Comparison: Healthy Control vs Exposed to HIV/HAART; T-test to detect differences between groups; Test type: Superiority or Other; p = 0.46, t-test, 2 sided

3. Secondary Outcome: Global Strain Rate
Description: Myocardial deformation (a measure of heart contractility) measured by speckel tracking echocardiography
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of full deformation
Arm/Group | Healthy Control | Exposed to HIV/HAART
Number analyzed (Participants) | 30 | 30
percentage of full deformation | -22.3 (3.2) | -21.1 (2.7)
Statistical Analysis 1: Comparison: Healthy Control vs Exposed to HIV/HAART; T-test to detect differences between groups; Test type: Superiority or Other; p = 0.13, t-test, 2 sided

4. Secondary Outcome: Systolic Myocardial Velocity During Systole (S')
Description: Systolic myocardial velocity during systole measured by tissue Doppler echocardiography
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Healthy Control | Exposed to HIV/HAART
Number analyzed (Participants) | 30 | 30
cm/s | 9.3 (1.1) | 9.1 (1.3)
Statistical Analysis 1: Comparison: Healthy Control vs Exposed to HIV/HAART; T-test to detect differences between groups; Test type: Superiority or Other; p = 0.59, t-test, 2 sided

5. Secondary Outcome: Early to Late Diastolic Filling Ratio
Description: Early to late diastolic filling ratio measured by tissue Doppler echocardiography
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ratio, unitless
Arm/Group | Healthy Control | Exposed to HIV/HAART
Number analyzed (Participants) | 30 | 30
ratio, unitless | 2.1 (0.5) | 1.8 (0.4)
Statistical Analysis 1: Comparison: Healthy Control vs Exposed to HIV/HAART; T-test to detect differences between groups; Test type: Superiority or Other; p = 0.09, t-test, 2 sided

6. Secondary Outcome: Myocardial Wall Velocity During Early Diastole
Description: Myocardial wall velocity during early diastolemeasured by tissue Doppler imaging
Time Frame: Baseline
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Healthy Control | Exposed to HIV/HAART
Number analyzed (Participants) | 30 | 30
cm/s | 16.3 (2.5) | 15.0 (2.2)
Statistical Analysis 1: Comparison: Healthy Control vs Exposed to HIV/HAART; T-test to detect differences between groups; Test type: Superiority or Other; p = 0.03, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Healthy Control: HIV-negative children born to healthy, HIV-negative women
  No adverse events
- Exposed to HIV/HAART: HIV-negative children exposed to HIV and HAART in utero
  No adverse events
Arm/Group | Healthy Control | Exposed to HIV/HAART
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No